CLINICAL TRIAL: NCT06875414
Title: Breast Cancer, Resilience, Quality of Life and Depression in Couples From Diagnosis to 24 Months Later: Prospective Pilot Study
Brief Title: Breast Cancer and Resilience in Couple
Acronym: resilience
Status: Recruiting | Type: Observational
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Principal Investigator, Silvia Takanen, Doctor Principal Investigator, Regina Elena Cancer Institute
Other Study IDs: RS1718/22(2657)
Record Dates: First submitted 2023-03-15; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Breast Neoplasms; Quality of Life
Keywords: breast cancer; quality of life; resilience; depression
MeSH Terms: conditions — Breast Neoplasms; Depression | interventions — Models, Nursing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Couple: The adaptation strategies that the couple uses
  Interventions: Behavioral: Nursing care model

INTERVENTIONS:
Behavioral: Nursing care model — Describe relation between resilience, quality of life and depression and marital adaptation in the population considered from diagnosis to 24 months later.

SUMMARY:
This is a prospective pilot study examining the couple's dyadic attitudes from diagnosis to 24 months later when one member is affected by illness and the adaptive strategies the couple employs when stressful events occur.

DETAILED DESCRIPTION:
The patients taking part in the study and their partners are examined from the time of the woman's breast cancer diagnosis up to 24 months later with the help of questionnaires and a focus group in order to understand the couple's coping strategies.

ELIGIBILITY:
INCLUSION CRITERIA:

* Woman diagnosed with stage 1, 2 or 3 breast cancer
* age> 18 years (patient and partner)
* The partner must have lived with the woman for at least 6 months at diagnosis and treatment
* Patients under treatment at the radiotherapy clinic
* Subjects available and able to answer questionnaires, interviews, and / or participate in focus groups
* Informed consent

EXCLUSION CRITERIA:

Cognitive deficits and / or inability to comply with the provisions of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of 40 couples with women affected by breast cancer who had lived together for at least six months before the diagnosis of breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-11-14 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2025-11-14 (Estimated)

PRIMARY OUTCOMES:
EORTC-QLQ C30 | 24 months
  The questionnaire EORTC-QLQ C30 (Kaasa, S., Bjordal, K., Aaronson, N.,1995) will evaluate the quality of life and will be administered to patients and their partners during a scheduled check-up visit at the Institute

SECONDARY OUTCOMES:
Marital Adjustment Test | 24 months
  Marital Adjustment Test (Locke and Wallace, 1959), this test validated in Italian, to investigate marital satisfaction, and will be administered to patients and their partners during a scheduled check-up visit at the Institute
PHQ-9 Scale | 24 months
  PHQ-9 Scale (Spitzer, Kroenke, Williams, 1999) validated in Italian, this questionnaire will be administered to patients and their partners during a scheduled check-up visit at the Institute to investigate psychological adjustment, in particular the presence of depression
Resilience Scale | 24 months
  Resilience Scale (Wagnild, G. M., & Young, H. M., 1993) validated in Italian, administered to patients and their partners during a scheduled check-up visit at the Institute to investigate resilience in adults.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Regina Elena National Cancer Institute, Roma, Rome, Italy

REFERENCES:
- [Result] Badger TA, Segrin C, Hepworth JT, Pasvogel A, Weihs K, Lopez AM. Telephone-delivered health education and interpersonal counseling improve quality of life for Latinas with breast cancer and their supportive partners. Psychooncology. 2013 May;22(5):1035-42. doi: 10.1002/pon.3101. Epub 2012 May 10. PMID 22573418
- [Result] Badr H, Krebs P. A systematic review and meta-analysis of psychosocial interventions for couples coping with cancer. Psychooncology. 2013 Aug;22(8):1688-704. doi: 10.1002/pon.3200. Epub 2012 Oct 9. PMID 23045191
- [Result] Belcher AJ, Laurenceau JP, Graber EC, Cohen LH, Dasch KB, Siegel SD. Daily support in couples coping with early stage breast cancer: maintaining intimacy during adversity. Health Psychol. 2011 Nov;30(6):665-73. doi: 10.1037/a0024705. Epub 2011 Aug 8. PMID 21823795
- [Result] Bigatti SM, Steiner JL, Makinabakan N, Hernandez AM, Johnston E, Storniolo AM. Matched and mismatched cognitive appraisals in patients with breast cancer and their partners: implications for psychological distress. Psychooncology. 2012 Nov;21(11):1229-36. doi: 10.1002/pon.2028. Epub 2011 Sep 1. PMID 21882286
- [Result] Brandao T, Schulz MS, Matos PM. Psychological intervention with couples coping with breast cancer: a systematic review. Psychol Health. 2014;29(5):491-516. doi: 10.1080/08870446.2013.859257. Epub 2013 Nov 27. PMID 24279379
- [Result] Christie KM, Meyerowitz BE, Stanton AL, Rowland JH, Ganz PA. Characteristics of breast cancer survivors that predict partners' participation in research. Ann Behav Med. 2013 Aug;46(1):107-13. doi: 10.1007/s12160-013-9477-7. PMID 23456213
- [Result] Dalton WT 3rd, Nelson DV, Brobst JB, Lindsay JE, Friedman LC. Psychosocial variables associated with husbands' adjustment three months following wives' diagnosis of breast cancer. J Cancer Educ. 2007 Winter;22(4):245-9. doi: 10.1007/BF03174124. PMID 18067437
- [Result] Duggleby W, Doell H, Cooper D, Thomas R, Ghosh S. The quality of life of male spouses of women with breast cancer: hope, self-efficacy, and perceptions of guilt. Cancer Nurs. 2014 Jan-Feb;37(1):E28-35. doi: 10.1097/NCC.0b013e31827ca807. PMID 23348665
- [Result] Fergus KD, Gray RE. Relationship vulnerabilities during breast cancer: patient and partner perspectives. Psychooncology. 2009 Dec;18(12):1311-22. doi: 10.1002/pon.1555. PMID 19353517
- [Result] Hoga LA, Mello DS, Dias AF. Psychosocial perspectives of the partners of breast cancer patients treated with a mastectomy: an analysis of personal narratives. Cancer Nurs. 2008 Jul-Aug;31(4):318-25. doi: 10.1097/01.NCC.0000305748.43367.1b. PMID 18600120
- [Result] Hubbard G, Menzies S, Flynn P, Adams S, Haseen F, Thomas I, Scanlon K, Reed L, Forbat L. Relational mechanisms and psychological outcomes in couples affected by breast cancer: a systematic narrative analysis of the literature. BMJ Support Palliat Care. 2013 Sep;3(3):309-17. doi: 10.1136/bmjspcare-2012-000274. Epub 2012 Oct 25. PMID 24644749
- [Result] Jun EY, Kim S, Chang SB, Oh K, Kang HS, Kang SS. The effect of a sexual life reframing program on marital intimacy, body image, and sexual function among breast cancer survivors. Cancer Nurs. 2011 Mar-Apr;34(2):142-9. doi: 10.1097/NCC.0b013e3181f1ab7a. PMID 20885305